CLINICAL TRIAL: NCT00096031
Title: Cetuximab As Second Line Therapy In Patients With Metastatic Esophageal Cancer - Phase II
Brief Title: S0415 Cetuximab in Treating Patients With Metastatic Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000391201; S0415 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): 250 mg/m^2 on days 1, 8, 15, and 22 of every 28-day cycle.
  Interventions: Biological: cetuximab

INTERVENTIONS:
Biological: cetuximab — 1 time Cetuximab 400mg/m2 IV over 120 minutes followed by weekly Cetuximab 250mg/m2 IV over 60 minutes.
  Other Names: Erbitux

SUMMARY:
RATIONALE: Biological therapies such as cetuximab may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well cetuximab works in treating patients with metastatic esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 6-month overall survival of patients with metastatic adenocarcinoma of the esophagus or gastroesophageal junction treated with cetuximab as second-line therapy.
* Determine the response rate (confirmed and unconfirmed, complete and partial), time to progression, and time to treatment failure in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Correlate, preliminarily, gene expression and germline polymorphism of enzymes and genes involved in the epidermal growth factor receptor pathway, DNA repair, and angiogenesis with time to progression, response, overall survival, toxic effects, and time to treatment failure in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours on day 1. Treatment repeats once weekly in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months until 3 years from the date of study registration.

PROJECTED ACCRUAL: A total of 30-55 patients will be accrued for this study within 6-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of 1 of the following sites:

  * Thoracic esophagus, located > 20 cm* from the incisors
  * Gastroesophageal junction, located ≤ 2 cm into the gastric cardia NOTE: *Tumors located < 26 cm from the incisors must be confirmed by bronchoscopy and negative cytology
* Disease confined to the esophagus and periesophageal soft tissue
* Metastatic disease
* Measurable disease by x-ray, scanning, or physical examination
* Received exactly 1 prior chemotherapy regimen for metastatic or recurrent disease

  * One prior adjuvant or neoadjuvant chemotherapy regimen allowed if administered at the time of initial diagnosis with localized disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine ≤ 1.5 times upper limit of normal

Other

* No prior allergic reaction to chimerized or murine monoclonal antibodies
* No evidence of human anti-mouse antibodies (HAMA)
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior cetuximab

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* At least 3 weeks since prior thoraco-abdominal surgery and recovered

Other

* No other prior therapy that specifically targets the epidermal growth factor pathway
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-10; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip J. Gold, MD, Study Chair — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus; Syma Iqbal, MD, Study Chair — University of Southern California
Locations (152):
- United States (152):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - John Smith, Jr. - Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Gold PJ, Goldman B, Iqbal S, et al.: Cetuximab as second-line therapy in patients with metastatic esophageal cancer: a phase II Southwest Oncology Group study. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-96, 2008.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab
Started | 63
Eligible | 57
Eligible and Began Protocol Therapy | 55
Completed | 0
Not Completed | 63
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 42
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 8
Not completed — Not protocol specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 61.2 [30.7 to 88.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 6 Months
Description: Time to death is measured from date of registration to date of death due to any cause.
Time Frame: every 3 weeks while on treatment, then every 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 55
percentage of participants | 36 [24 to 50]

2. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is measured from date of registration to date of first observation of progressive disease, death due to any cause, symptomatic deterioration, or early discontinuation of treatment. Progressive disease is defined as one or more of the following: 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is defined as global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: every 3 weeks while on treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 55
months | 1.8 [1.7 to 1.9]

3. Secondary Outcome: Time to Progression
Description: Progression free survival is measured from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact. Progressive disease is defined as one or more of the following: 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is defined as global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: every 3 weeks while on treatment, then every 3 months for 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 55
months | 1.8 [1.7 to 1.9]

ADVERSE EVENTS:
Time Frame: After every 28 days while on treatment
Description: Standard AE form
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=55)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=55)
Hemoglobin (Blood and lymphatic system disorders) | 25
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 23
Pain - Abdomen NOS (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 10
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34
Rigors/chills (General disorders) | 3
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 4
Alkaline phosphatase (Investigations) | 7
Bilirubin (hyperbilirubinemia) (Investigations) | 4
Leukocytes (total WBC) (Investigations) | 3
Platelets (Investigations) | 3
Weight loss (Investigations) | 6
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 11
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4
Pain - Head/headache (Nervous system disorders) | 8
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 9
Nail changes (Skin and subcutaneous tissue disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No